CLINICAL TRIAL: NCT02033525
Title: A Phase I-IIa Safety and Efficacy Pilot Clinical Trial of Intraarticular Administration of Autologous Mesenchymal Cells for Meniscus Injury
Brief Title: Mesenchymal Stromal Cells for Degenerative Meniscus Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Collaborators: Hospital Universitari Quirón Dexeus (Unknown); Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XCEL-MEN-01; 2011-006270-13 (EudraCT Number)
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Chronic Meniscal Injury
Keywords: Chronic Meniscal Injury; Degenerative meniscus; Meniscus injury; Meniscal injury; Mesenchymal stromal cells; Mesenchymal stem cells; Advanced Therapy; Bone marrow
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XCEL-M-ALPHA and standard rehabilitation (Experimental): Intraarticular administration of XCEL-M-ALPHA followed by standard rehabilitation program
  Interventions: Drug: XCEL-M-ALPHA and standard rehabilitation
- standard rehabilitation (Active Comparator): Standard rehabilitation program
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Drug: XCEL-M-ALPHA and standard rehabilitation — Intraarticular infusion of autologous bone marrow derived ex vivo expanded mesenchymal stromal cells produced at Xcelia (Advanced Therapies Division of the Blood and Tissue Bank)
  Other Names: XCEL-M-ALPHA
  Arms: XCEL-M-ALPHA and standard rehabilitation
Other: Rehabilitation — Standard rehabilitation program
  Arms: standard rehabilitation

SUMMARY:
The present proposal has the objective to assess whether the addition of autologous ex vivo expanded mesenchymal stromal cells (XCEL-M-ALPHA) to the conventional meniscal injury rehabilitation program is contributing in creating the proper healing environment for the meniscus repair. For this purpose, 20 patients will be randomized (10 per group) to one of the two treatment arms (rehabilitation + xcel-m-alpha or rehabilitation alone) . The conduction of this clinical trial will, in addition of having the aim of improving the patient's quality of life, contribute to consolidate an emerging new type of therapy which is still under development.

DETAILED DESCRIPTION:
This is a prospective, unicentric, randomized, open-label, single-dose, two-arm, blinded assessor pilot study in which 20 patients with degenerative meniscus injury grade 3 (Crues et al.) will enter the study with the primary objective of assessing the efficacy of the treatment by VAS of pain at 12 month. Secondary objectives are to evaluate the safety and efficacy through imaging procedures and clinical questionnaires (IKDC, KOOS, Lysholm and SF-36.

Patients will be randomized to one of the two treatment arms (XCEL-M-ALPHA and standard rehabilitation program or standard rehabilitation program alone). Thereafter, patients will be followed for 12 months.

Imaging assessment will be performed by an independent blinded radiologist.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 40 and 60 years of age
* Degenerative meniscus injury grade 3 (Crues et al.)
* Indication of conservative treatment
* Normal alignment of the knee (between 3º varus and 10 º valgus)
* Patient is able to follow a rehabilitation program
* Informed consent given by the patient in writing
* Patient is able to understand the trial.

Exclusion Criteria:

* Traumatic meniscus injury
* Surgical intervention to the affected knee
* Local or systemic infection
* Intraarticular treatment of the affected knee with steroids or hyaluronic acid within the past 3 months
* Significant abnormal laboratory tests that contraindicates participation in the trial.
* Pregnant women or intend to become pregnant or breast-feeding
* Neoplastic process within the previous 5 years or without complete remission.
* The patient is wearing a pacemaker, allergy to contrast, severe renal insufficiency or any other condition that contraindicates the magnetic resonance using contrast.
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria
* Legally dependant patient.
* The patient does not accept to be followed-up for a period that could exceed the clinical trial length

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
VAS for pain | 12 month
  Visual analogue scale (VAS) for pain at 12 month follow-up.

SECONDARY OUTCOMES:
Safety | 12 month
  Safety will be assessed by collecting adverse events, physical exam, laboratory tests, and vital signs.
Efficacy by MRI | 6 and 12 month
  Efficacy will be assessed by qualitative and quantitative changes of the meniscus and articular cartilage by imaging procedures (MRI) at 6 and 12 month follow-up.
VAS for pain | 1, 3 and 6 month
  Visual analogue scale (VAS) for pain at 1, 3 and 6 month follow-up.
Efficacy by clinical questionnaires | 3, 6 and 12 month
  IKDC, KOOS and Lysholm functionality test and SF-36 quality of life at 3, 6 and 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Joan Carles Monllau, MD, PhD, Principal Investigator — ICATME-Hospital Quiron Dexeus
Locations (1):
- ICATME-Hospital Quiron Dexeus, Barcelona, Spain

REFERENCES:
- See also: Fundación ICATME (Spanish only) — http://www.icatme.com/